CLINICAL TRIAL: NCT02054286
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase I/II Trial to Compare the Safety, Tolerability and Immunogenicity of the Therapeutic THV01 Vaccination at 5.10E+6 TU (Transducing Unit) , 5.10E+7 TU (Transducing Unit) or 5.10E+8 TU (Transducing Unit) Doses to Placebo in HIV-1 Clade B Infected Patients Under Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety, Tolerability and Immunogenicity Induced by the THV01 Treatment in Patients Infected With HIV-1 Clade B and Treated With Highly Active Antiretroviral Therapy (HAART).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theravectys S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THV01-11-01
Record Dates: First submitted 2014-02-01; First posted 2014-02-04 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: THV01 (5.10E+6 TU) or Placebo (Experimental): 5.10E+6 TU (transducing unit) of THV01-1 (Week 0) OR matching placebo; 5.10E+6 TU (transducing unit) of THV01-2 (Week 8) OR matching placebo
  Interventions: Biological: THV01-1; Biological: THV01-2; Biological: Placebo
- Group 2: THV01 (5.10E+7 TU) or Placebo (Experimental): 5.10E+7 TU (transducing unit) of THV01-1 (Week 0) OR matching placebo; 5.10E+7 TU (transducing unit) of THV01-2 (Week 8) OR matching placebo
  Interventions: Biological: THV01-1; Biological: THV01-2; Biological: Placebo
- Group 3: THV01 (5.10E+8 TU) or Placebo (Experimental): 5.10E+8 TU (transducing unit) of THV01-1 (Week 0) OR matching placebo; 5.10E+8 TU (transducing unit) of THV01-2 (Week 8) OR matching placebo
  Interventions: Biological: THV01-1; Biological: THV01-2; Biological: Placebo

INTERVENTIONS:
Biological: THV01-1 — Intramuscular injection of THV01-1 (week 0)
  Other Names: lentiviral vector ancoding an HIV antigen
Biological: THV01-2 — Intramuscular injection of THV01-2 (week 8)
  Other Names: lentiviral vector encoding an HIV antigen
Biological: Placebo — Intramuscular injection of placebo matching THV01-1 and THV01-2
  Other Names: Placebo matching THV01-1 and THV01-2

SUMMARY:
The objectives of this Phase I/II trial is to evaluate the safety, tolerability and immunogenicity of THV01 compared to placebo in HIV-1 infected patients on HAART (highly active antiretroviral therapies).

THV01 is composed of two vaccines that derived from the HIV (human immunodeficiency virus): lentiviral vectors. They are non-replicative and not infectious. They will be injected intramuscularly, eight weeks apart. Three doses will be assessed and compared to placebo.

Eligible patients must have an undetectable viral load and must be treated by HAART for more than 12 months. They will be randomly allocated to one of the study group and will receive the experimental drugs at one of the three doses or a matching placebo.

Their anti-HIV treatment will be alleviated around each experimental drugs' administration to enable THV01 efficacy. HAART will be resumed one week after the second injection. 15 weeks after resumption, HAART will be interrupted. Patients will then be monitored every 2 weeks for CD4+ T cell counts and viral load as well as for thorough assessment of the elicited immune response. Stringent anti-HIV treatments resumption criteria have been implemented, based on the CD4+ T cell counts and the viral load.

38 patients were enrolled in THV01-11-01 study and received the 2 injections.

A long-term follow-up of all enrolled patients will be performed for 5 years post-prime administration. This will provide additional data on the safety and the potential long-term risks/benefits associated with THV01.

The final study report will be written after the last patient last visit in the long-term follow-up.

DETAILED DESCRIPTION:
This Phase I/II is a randomized, double-blind and placebo controlled study to assess safety, tolerability and immunogenicity of THV01 at three doses in patients infected with the HIV-1 clade B currently on HAART (highly active antiretroviral therapies).

THV01 involves two intramuscular injections, consisting of the THV01-1 and THV01-2 lentiviral vectors, to be administered intramuscularly eight weeks apart. These lentiviral vectors are non-replicative and self-inactivating. Both encode the same HIV antigen.

36 patients were planned to be enrolled. They must be HIV-1 (clade B) infected patients, treated by HAART for more than 12 months and with an undetectable viral load.

Patients will be randomly allocated to one of the groups:

* Group 1: patients will receive the THV01-1 and THV01-2 vaccines at 5.10E+6 TU (transducing unit) or placebo;
* Group 2: patients will receive the THV01-1 and THV01-2 vaccines at 5.10E+7 TU (transducing unit) or placebo;
* Group 3: patients will receive the THV01-1 and THV01-2 vaccines at 5.10E+8 TU (transducing unit) or placebo.

Hence, twelve patients will be randomized in blocks of 4 in a 3:1 ratio (vaccine:placebo) for each dose.

Experimental drugs' injection will occur at Week 0 and Week 8. HAART will be alleviated for all patients during this "vaccination phase" to enable efficient transduction of the host cells by the lentiviral vectors. Initial HAART will be resumed at Week 9.

Starting on Week 24, HAART will be interrupted. Patients will then be monitored on a very stringent rhythm. HAART resumption criteria based on the CD4+ T cell counts and the viral load have been implemented to guaranty safety of all enrolled patients.

38 patients were enrolled in THV01-11-01 study and received the 2 injections.

A long-term follow-up of all enrolled patients will be performed for 5 years after the administration of THV01-1. During this follow-up, three visits are planned per year, during which blood will be sampled. This will provide data on the long-term safety of THV01 and the potential long-term risks/benefits associated with THV01.

ELIGIBILITY:
Inclusion criteria

* Patients infected with clade B HIV-1;
* Confirmation of a Gag clade B genotyping performed at screening;
* Patient must be treated by a triple agents therapy for more than 12 months at baseline: this triple agents therapy should encompasses two (2) nucleosidic reverse transcriptase inhibitors plus one (1) boosted protease inhibitor, or two (2) nucleosidic reverse transcriptase inhibitors plus one (1) non nucleosidic reverse transcriptase inhibitor;
* Patients must be treated for more than 60 days at baseline by two (2) nucleosidic reverse transcriptase inhibitors plus a ritonavir boosted protease inhibitor treatment among darunavir+ritonavir or lopinavir+ritonavir;
* Patients' HIV plasma viral load ≤150,000 copies mL-1 at any monitoring time (apart measurement during primo-infection if recorded);
* Patients with HIV plasma viral load persistently ≤ 50 copies mL-1 during the 12 months prior to screening;
* Patients' CD4+ T cells count ≥ 300 cells per mm3 at any time since diagnosis;
* Patient's CD4+ T cells count < 500 cells per mm3 at least once from diagnosis to initiation of antiretroviral treatment;
* Patients with CD4+ T cells count ≥ 600 cells per mm3 at baseline;
* Man or woman aged 18-55 years;

Exclusion Criteria

* HIV-2 infection;
* Patient treated by HIV entry of fusion inhibitors;
* Patient treated by HIV integrase inhibitors;
* Patient displaying any HIV protease inhibitor resistance mutation as listed in the current version of the HIV drug resistance database (Stanford University);
* Patient having undergone virological failure as defined by a viral load ≥ 500 copies mL-1 confirmed by a second measure, since initiation of treatment;
* More than 2 blips with viral load comprised between 50 and 500 copies mL-1 during the 12 months prior inclusion;
* History of an AIDS-defining clinical illness;
* Concomitant AIDS-related opportunistic disease;
* History of allergic disease, anaphylaxis or reactions likely to be triggered or exacerbated by any component of the vaccine such as lactose;
* Acute or chronic infectious disease other than AIDS (include but not limited to viral hepatitis such as hepatitis B and hepatitis C, active tuberculosis, active syphilis, HTLV-1, HTLV-2);
* Acute, chronic or history of clinically relevant pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable CNS pathology, angina or cardiac arrhythmias, or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
* Severe hepatic impairment;
* Serious dyslipidaemia;
* Severe disorders of blood coagulation;
* Known or suspected allergy to egg phospholipids, soy proteins and/or peanut;
* Acute, chronic or history of immunodeficiency or autoimmune disease other than HIV infection;
* Unstable asthma (defined as sudden acute attacks occurring in less than three hours without an obvious trigger, hospitalisation for asthma in the last two years); food or wine induced asthma;
* History of malignancy unless there has been surgical excision that is considered to have achieved cure;
* Active malignancy that may require chemotherapy or radiation therapy;
* Seizure disorder or any history of prior seizure;
* Subjects planning to receive a prophylactic or therapeutic vaccination during the study except Influenza immunization;
* Subjects who have received any vaccination for the 3 months prior the first injection;
* Subjects having an infective exacerbation as defined as a requirement of inhaled, oral, or intravenous antibiotics at W-2 or later;
* Serious illness requiring systemic treatment and/or hospitalization within 7 days prior to baseline;
* Pregnant or breast-feeding woman;
* Any contraindication of intramuscular injection;
* Active drug or alcohol abuse or dependence;
* Any condition, which in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From Week 0 to Week 24
  Occurrence of at least one grade 3 or higher adverse event including signs/symptoms, laboratory toxicities and/or clinical events possibly, probably or definitely related to study treatment.

SECONDARY OUTCOMES:
Safety and tolerability | From baseline to Week 88 (or early termination).
  Occurrence of at least one grade 3 or higher adverse event including signs/symptoms, laboratory toxicities and/or clinical events possibly, probably or definitely related to study treatment.
Immunogenicity | From baseline to Week 88 (or early termination).
  Monitoring the cellular immune response by treatment group versus placebo.

OTHER OUTCOMES:
HIV reservoir (HIV total DNA) | From baseline to five years after the prime injection.
  Evaluation of HIV reservoir by treatment group versus placebo.
Long term safety | From Week 88 to five years after the prime injection.
  Occurrence of any SAE (serious adverse event) suspected to be related to IMP.

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Pr, Principal Investigator — CIC Cochin-Pasteur; Hôpital Cochin; Paris
Locations (11):
- Belgium (2):
  - CHU Saint-Pierre, Brussels
  - CHU Liège, Liège
- France (9):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Croix-Rousse, Lyon
  - Hôpital Saint-Louis, Paris
  - CIC Cochin-Pasteur; Hôpital Cochin, Paris
  - CHU Rennes, Rennes
  - Hôpital Nord, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - Hôpital Purpan, Toulouse